CLINICAL TRIAL: NCT04707651
Title: Formula Diet Treatment for Weight Reduction in NASH Patients.
Brief Title: Formula Diet Treatment for NASH Patients.
Acronym: NASH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Responsible Party: Principal Investigator, Stephan Martin, Principal investigator, West German Center of Diabetes and Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NASH
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Steatohepatitis, Nonalcoholic
Keywords: overweight; fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Fatty Liver | interventions — Food, Formulated

STUDY DESIGN:
Intervention Model Description: Lifestyle intervention including formula diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention (Experimental): Nutrition advices and formula diet
  Interventions: Dietary Supplement: Formula diet

INTERVENTIONS:
Dietary Supplement: Formula diet — Formula diet for 12 weeks

SUMMARY:
Non-alcoholic steatohepatitis (NASH) - also called fatty liver - is medically a serious problem because the liver tissue becomes fatty and stiff, and inflammatory reactions occur. This increases the risk of liver fibrosis (= scarring of the liver), liver cirrhosis (= shrunken liver), a liver tumor or death. So far there is no recognized treatment option for this disease. However, there is evidence that a lifestyle change based on a reduced carbohydrate diet, more exercise and a significant weight loss that can improve NASH.

DETAILED DESCRIPTION:
Outpatients with NASH will be included into this lifestyle intervention study. Patients will get nutritional advices and a formula diet for 12 weeks. Clinical visits will take place at baseline, after 4, 12 and after 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25 kg/qm

Exclusion Criteria:

* history of drug or alcohol abuse
* acute or chronic diseases (except type 2 diabetes)
* pregnancy or breast feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
degree of steatosis | 12 weeks
  degree of steatosis in decibels per meter (dB/m) measured by Controlled Attenuation Parameter (CAP) estimation

SECONDARY OUTCOMES:
degree of steatosis | 52 weeks
  degree of steatosis in decibels per meter (dB/m) measured by Controlled Attenuation Parameter (CAP) estimation
degree of fibrosis | 12 weeks and 52 weeks
  degree of fibrosis in meter per second (m/s) measured by Acoustic Radiation Force Impulse (ARFI) elastography
fat mass | 12 weeks and 52 weeks
  fatt mass in kilogram (kg) measured by Bioelectrical Impedance Analysis (BIA)
Glutamate Pyruvate Transaminase (GPT) | 12 weeks and 52 weeks
  Glutamate Pyruvate Transaminase in units/litre (U/L)
Gamma-glutamyltransferase (GGT) | 12 weeks and 52 weeks
  Gamma-glutamyltransferase in units/litre (U/L)
insulin | 12 weeks and 52 weeks
  insulin in micro units per millilitre (µU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West-German Centre of Diabetes and Health
Locations (2):
- Germany (2):
  - Düsseldorf Catholic Hospital Group, Düsseldorf
  - Praxis Prof. Erhardt, Wuppertal